CLINICAL TRIAL: NCT06761781
Title: Augmented Reality for Stroke Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/01997 Abrish Habib
Record Dates: First submitted 2025-01-01; First posted 2025-01-07 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Stroke/Brain Attack
Keywords: Stroke rehabilitation; Augmented reality; Balance; motor function
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Augmented Reality Training (Experimental): Augmented reality training to Experimental group
  Interventions: Other: Augmented Reality
- Traditional Treatment (Active Comparator): Task based training to the Control Group
  Interventions: Other: Traditional Training

INTERVENTIONS:
Other: Augmented Reality — Each participant will receive a standard trial consisting of 20 training sessions (2-5 sessions per week, 120 min per session) in consecutive 4-10 weeks. Each session will consist of 2-10 exercises selected by the trainer from a pool of 46 exercises. The selected exercises will be tailored based on the participant's condition and progress. The exercise pool will be designed as comprehensively as possible to cover the upper limb (22 exercises and lower limb (7 exercises) motor functions, balance ability (11 exercises), or/and coordination (6 exercises).
  Each exercise with a duration ranging from 3 to 23 min, and will be determined by a set of parameters that can be adjusted to the individuals dynamically according to the participant's performance.
  Arms: Augmented Reality Training
Other: Traditional Training — Each participant will receive a Traditional training based on Task oriented training consisting of 20 training sessions (2-5 sessions per week, 120 min per session) in consecutive 4-10 weeks. Exercises will be tailored based on the participant's condition and progress. The exercises will cover the upper limb, lower limb, motor functions, balance ability and coordination.
  Arms: Traditional Treatment

SUMMARY:
The study aims to determine the effectiveness of Augmented reality on motor function, balance, and functional ambulation in stroke patients.

DETAILED DESCRIPTION:
The study aims to determine the effectiveness of Augmented reality on motor function, balance, and functional ambulation in stroke patients. The emerging technology of Augmented Reality (AR), has been validated as a promising way to assist the rehabilitation training in Stroke patients. The purpose of this study is to investigate the feasibility of the AR rehabilitation system in a real-world setting. The following questions will be addressed by the present study: (a) How the Augmented reality effects motor function, balance, and functional ambulation in stroke patients? (b) how much and what types of manpower can be saved while maintaining the efficacy of training with the assistance of the AR rehabilitation? (c) how can the contact rate be reduced with the AR training? (d) how do therapists/patients experience the AR training?

ELIGIBILITY:
Inclusion Criteria:

Participants falling in this category would be recruited into the study.

1. age between 18 to 90 years who are diagnosed with ischemic brain injury, intracerebral hemorrhage shown by magnetic resonance imaging, or computed tomography after the onset of stroke;
2. with motor impairment in the upper limb, lower limb, and/or balance;
3. have no or mild spasticity on the lower limb or upper limb assessed by Modified Ashworth Scale (MAS ≤ 2); and
4. have sufficient cognition to follow the instructions provided by the therapists and the computer.

Exclusion Criteria:

Participants fall in this category would be excluded of the study.

1. any additional medical or psychological condition that would affect their ability to comply with the study protocol, e.g., a significant orthopedic or chronic pain condition, major post-stroke depression, epilepsy, artificial cardiac pacemaker/joint;
2. have severe shoulder/arm or hip/knee contracture/ pain and;
3. Pregnant women.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2024-12-31 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment Upper Extremity and Lower Extremity (FMA-UE and FMA-LE); | 10 weeks
  The cumulative test score for all components is 226 with availability of specific subtest scores (e.g., UE maximum score is 66, LE score 34; balance score 14). This instrument has good construct validity and high reliability (r 0.99) for determining motor function.
Berg Balance Scale (BBS); | 10 weeks
  The Berg Balance Scale (BBS) is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function and takes approximately 20 minutes to complete.
Functional Ambulation Category (FAC) | 10 weeks
  The Functional Ambulation Categories (FAC) is a 6-point functional walking test that evaluates ambulation ability, determining how much human support the patient requires when walking, regardless of whether or not they use a personal assistive device. The FAC is a quick visual measurement of walking, is simple to use, easy to interpret. The test has good interrater reliability (κ=.72) and excellent test-retest reliability (k=.950).

SECONDARY OUTCOMES:
Quality of life (QOL): physical and mental health using the 12-Item Short Form Health Survey (SF 12v2) | 10 weeks
  The 12-Item Short Form Health Survey (SF-12v2) is a validated questionnaire widely used to assess health-related quality of life (HRQOL) focusing on both physical and mental health dimensions. The SF-12v2 consists of 12 questions that cover eight domains of health, leading to two primary summary scores:
  Physical Component Summary (PCS) and Mental Component Summary (MCS).The SF-12v2 exhibits high internal consistency, with Cronbach's alpha coefficients typically exceeding 0.80 for both the PCS and MCS components.
User experience (UX) using questionnaires (designed based on UEQ-S) | 10 weeks
  User Experience (UX) encompasses all aspects of the end-user's interaction with a company, its services, and its products. To systematically evaluate UX, particularly in digital products. The UEQ-S consists of 8 items that are grouped into 6 key dimensions of user experience.The UEQ-S shows high internal consistency, with Cronbach's alpha values generally exceeding 0.70 for the various dimensions, ensuring that the items within each dimension measure a coherent aspect of user experience.
Activities of Daily Living (ADL) using the Barthel Index (BI) | 10 weeks
  The Barthel Index (BI) is a widely recognized tool for assessing an individual's ability to perform Activities of Daily Living (ADLs). It evaluates the extent to which individuals can maintain self-care and functional independence. The Barthel Index consists of 10 items.Each item is scored based on the level of independence demonstrated, with total scores ranging from 0 to 100. Higher scores indicate greater independence in performing daily activities. The Barthel Index exhibits high internal consistency, with Cronbach's alpha values typically above 0.80.

CONTACTS AND LOCATIONS:
Overall Officials: Arshad Nawaz Malik, PhD Rehab, Principal Investigator — Riphah International University; Abrish Habib Abbasi, PhD* Rehab, Principal Investigator — Riphah International University; Mirza Obaid Baig, MS-NMPT, Principal Investigator — Riphah International University
Locations (1):
- Railway General Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No